CLINICAL TRIAL: NCT04472338
Title: PATROL: Prostate Cancer Screening for People AT Genetic Risk FOr Aggressive Disease
Brief Title: Prostate Cancer Screening for People at Genetic Risk for Aggressive Disease, PATROL Study
Status: Recruiting | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Canary Foundation (Other); CureBRCA (Unknown)
Responsible Party: Sponsor
Other Study IDs: RG1004195; NCI-2020-04602 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 8760 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1004195 (Other: Fred Hutch/University of Washington Cancer Consortium); P50CA097186 (NIH)
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-09

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening (biospecimen collection): Participants undergo collection of blood, urine, and/or tissue samples every 12 months, when any biopsy occurs, and if relevant, at time of curative therapy and 12 months after completion of curative therapy.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood, urine, and/or tissue samples
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This study investigates ways to detect prostate cancer earlier in people at genetic risk for disease that forms, grows, or spreads quickly (aggressive). Studying samples of blood, urine, and/or tissue in the laboratory may help doctors further understand the genetics of prostate cancer and help identify ways to detect cancer earlier, thereby improving treatment and methods of early detection in the future.

DETAILED DESCRIPTION:
OUTLINE:

Participants undergo collection of blood, urine, and/or tissue samples every 6-12 months, when any biopsy occurs, and if relevant, at time of curative therapy and 3-9 months after completion of curative therapy for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* People with prostates ≥40 years of age
* Documented germline pathogenic variant in known or suspected genes associated with prostate cancer risk.

Exclusion Criteria:

* Prior diagnosis of prostate cancer
* Medical contraindication to any of the study procedures (e.g., prostate biopsy)
* For all cancer types except non-melanoma skin cancer, any cancer treatment with curative intent within the past 12 months (e.g., surgery, radiation, chemotherapy, immunotherapy)
* Prior or concurrent participation in an interventional clinical trial aimed at preventing cancer for people with germline variants associated with increased prostate cancer risk
* Unable to provide written informed consent
* Unable or unwilling to complete clinical care and study procedures as indicated by the study protocol.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — People with prostates
Study Population: Germline carriers of pathogenic or likely pathogenic mutations in genes associated with increased risk of prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Positive predictive values (PPVs) of age-based prostate specific antigen (PSA) thresholds | Up to 10 years
  To estimate PPVs of age-based PSA thresholds for biopsy referral in this patient population, will first fit a logistic regression model to estimate the odds that biopsy leads to a prostate cancer diagnosis. The regression will have a binary indicator of prostate cancer diagnosis as the response variable, patient age at biopsy (categorized as < 50, 50-59, or >= 60 years to correspond to the age-based PSA thresholds) as a fixed effect, and a unique patient identifier as a random effect to account for possibly repeated biopsies. Will then convert the estimated odds that biopsy leads to a prostate cancer diagnosis within each age category into corresponding probabilities of this outcome-i.e., PPV point estimates and associated 95% confidence intervals-using the inverse logit function.

CONTACTS AND LOCATIONS:
Overall Officials: Heather H. Cheng, MD, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - University of California, San Francisco, San Francisco, California
  - Northwestern, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - OHSU Knight Cancer Institute, Portland, Oregon
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No